CLINICAL TRIAL: NCT04913636
Title: A Pilot Clinical Study to Determine the Effect Denture Gel Has on the Prevention of Gum Abrasions
Brief Title: Assessing Effects of a Denture Gel on Gum Abrasions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020089
Record Dates: First submitted 2021-05-28; First posted 2021-06-04 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Gum Injury

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Test Group (Experimental)
  Interventions: Device: Treatment Gel
- Control Group (Sham Comparator)
  Interventions: Other: Sham Control

INTERVENTIONS:
Device: Treatment Gel — In the evening subjects will perform their regular denture cleaning routine. They will be instructed to sleep without dentures. Subjects will rinse out their mouth with water (if subjects brush their oral mucosa with brush, they will be allowed to continue doing so) and apply the gel to their mucosa where they normally wear upper or lower denture.
  Arms: Test Group
Other: Sham Control — Subjects will perform their regular denture cleaning routine.
  Arms: Control Group

SUMMARY:
This is a parallel design study. Up to 40 subjects with a full mandibular and full maxillary dentures will be enrolled into the study. Subjects will use their current denture care +/- a treatment gel for 4 weeks. Subjects will have an Oral Soft Tissue exam, a Mucosa Condition Assessment, and a Pre-Gum Abrasion Evaluation followed by a peanut challenge and then have a Post-Gum Abrasion Evaluation at designated timepoints.

DETAILED DESCRIPTION:
This is a single center, two-treatment, parallel design study. Up to 40 subjects will be enrolled with a full mandibular and full maxillary denture with a history of food related abrasions.

At each visit, an Oral Soft Tissue exam, a Mucosa Condition Assessment and a Gum Abrasion Evaluation will be performed. At Baseline, the subjects will be randomized to a treatment group. At Baseline, Week 2, and Week 4 subjects will be asked to eat 20 grams of peanuts 4 times for a total consumption of 80 g of peanuts (subjects will be permitted to take breaks if needed and drink small sips of water). Following the peanut challenge, a licensed dental professional will re-evaluate the number and size of abrasions. Subjects will receive a consumer questionnaire to complete as well prior to the Baseline, Week 2, and Week 4 assessments.

ELIGIBILITY:
Inclusion Criteria:

In order to be included in the study, each subject must:

* Be 18 years of age;
* Read, sign, and receive a copy of the Informed Consent prior to initiation of study procedures;
* Have a full maxillary and mandibular denture and wear on a daily basis;
* Have a history of food particles getting under their full denture and causing gum irritation;
* Are willing to abstain from eating at least four hours prior to the visits;
* Are willing to eat 4 X 20 grams of peanuts three times (Baseline, Week 2 and Week 4) without denture adhesive;
* Clean their dentures on a daily basis;
* Agree not to change their regular denture cleaning routine;
* Agree to abstain from using denture adhesive during the study;
* Agree to not participate in any other oral/dental product studies during the study.

Exclusion Criteria:

* Exhibit evidence of obvious oral pathology, as determined by the Study Dentist, as a result of a mandatory OST examination on the first day of the study;
* Are allergic to any of the ingredients contained in the study product gel;
* Are allergic to peanuts;
* Wear dentures overnight;
* Are insulin-dependent and/or have any health condition(s) which would prevent compliance with study procedures;
* Are routinely using denture adhesive;
* Present with any disease or conditions that could be expected to increase their susceptibility to gum abrasion (like diabetes or xerostomia); or
* Present with any disease or conditions that could be expected to interfere with examination procedures or the subject's safe completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Group | Control Group
Started | 18 | 20
Completed | 18 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Group | Control Group | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (12.39) | 64.4 (12.55) | 65.0 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 15 | 18 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Post-Peanut Gum Abrasion Evaluation (number) [Median (Standard Deviation); unit: number of abrasions] — Population: Subject dropped from experimental leg
  number of abrasions
    number analyzed (Participants) | 17 | 20 | 37
    (all) | 5.18 (3.729) | 3.85 (2.700) | 4.46 (3.237)
Post-Peanut Challenge Evaluation (size) [Mean (Standard Deviation); unit: mm] — Population: Subject dropped from experimental leg
  mm
    number analyzed (Participants) | 17 | 20 | 37
    (all) | 9.85 (7.678) | 5.95 (5.275) | 7.74 (6.690)

OUTCOME MEASURES:

1. Primary Outcome: Abrasion Assessment (Number)
Description: The total number of abrasions pre-food challenge
Time Frame: Day 3
Measure: Mean (Standard Error); unit: number of abrasions
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 16 | 20
number of abrasions | 3.65 (.518) | 4.11 (.461)

2. Primary Outcome: Abrasion Assessment (Size)
Description: The average size/area (in mm) of the total number of abrasions pre-food challenge
Time Frame: Day 3
Measure: Mean (Standard Error); unit: mm
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 16 | 20
mm | 6.77 (.731) | 7.24 (.653)

3. Primary Outcome: Abrasion Assessment (Number)
Description: The total number of abrasions pre-food challenge
Time Frame: Day 6
Measure: Mean (Standard Error); unit: number of abrasions
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 15 | 18
number of abrasions | 2.25 (.731) | 3.66 (.654)

4. Primary Outcome: Abrasion Assessment (Number)
Description: The total number of abrasions pre-food challenge
Time Frame: Week 2
Measure: Mean (Standard Error); unit: number of abrasions
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 15 | 18
number of abrasions | 2.23 (.688) | 2.48 (.627)

5. Primary Outcome: Abrasion Assessment (Number)
Description: The total number of abrasions pre-food challenge
Time Frame: Week 4
Measure: Mean (Standard Error); unit: number of abrasions
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 15 | 18
number of abrasions | 0.98 (.316) | 1.74 (.288)

6. Primary Outcome: Abrasion Assessment (Size)
Description: The average size/area (in mm) of the total number of abrasions pre-food challenge
Time Frame: Day 6
Measure: Mean (Standard Error); unit: mm
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 15 | 18
mm | 2.67 (1.079) | 5.58 (.981)

7. Primary Outcome: Abrasion Assessment (Size)
Description: The average size/area (in mm) of the total number of abrasions pre-food challenge
Time Frame: Week 2
Measure: Mean (Standard Error); unit: mm
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 15 | 18
mm | 3.18 (.523) | 2.20 (.476)

8. Primary Outcome: Abrasion Assessment (Size)
Description: The average size/area (in mm) of the total number of abrasions pre-food challenge
Time Frame: Week 4
Measure: Mean (Standard Error); unit: mm
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 15 | 18
mm | 2.15 (.647) | 3.39 (.588)

9. Primary Outcome: Mucosal Assessment
Description: The mucosal region under the denture was assessed with one score per arch (two total arches) each arch is scored ranging from 0(better) - 3(worse). The scores are then summed for a total score.
  The scale is measured as follows: 0 = pink firm tissue absent of redness and inflammation; 1 = mild redness or inflammation - slight change in color and little change in texture; 2 = moderate redness and/or inflammation - moderate glazing, redness, edema and hypertrophy 3 = severe redness and/or inflammation - marked redness and hypertrophy.
Time Frame: Day 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 16 | 20
units on a scale | .97 (.048) | 1.04 (.043)

10. Primary Outcome: Mucosal Assessment
Description: as for outcome 9
Time Frame: Day 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 15 | 18
units on a scale | .77 (.049) | 1.05 (.044)

11. Primary Outcome: Mucosal Assessment
Description: as for outcome 9
Time Frame: Week 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 15 | 18
units on a scale | .70 (.062) | 1.03 (.056)

12. Primary Outcome: Mucosal Assessment
Description: as for outcome 9
Time Frame: Week 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 15 | 18
units on a scale | .60 (.062) | 1.06 (.056)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for all four weeks of study duration.
Arm/Group | Test Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 2/18 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Group (N=18) | Control Group (N=20)
Mouth Ulceration (Gastrointestinal disorders) | 2 (4) | 0 (0)
Desquamation Oral (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI should disclose plans to sponsor prior to public release.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT04913636/Prot_SAP_000.pdf